CLINICAL TRIAL: NCT05440461
Title: Analysis of Psychometric Properties and Cultural Adaptation of Urdu Version of Oxford Knee Score in Patients With Knee Osteoarthritis
Brief Title: Reliability and Validity Study of Urdu Version of Oxford Knee Score in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/FSD/0290
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: Oxford Knee Score; Urdu Version; Reliability; Validity; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* To translate the Oxford knee score into Urdu language
* To evaluate the reliability and validity of Urdu Version of Oxford knee score for accessing pain and physical function in patients with knee osteoarthritis.
* To evaluate the correlation of Oxford knee score with Western Ontario McMaster universities osteoarthritis index and International Knee Documentation Committee

DETAILED DESCRIPTION:
The original English version of Oxford Knee Score will be translated and culturally adapted as per previous recommendation. In patients with knee osteoarthritis, Urdu Version of Oxford Knee Score will be distributed among 100 participants choose a convenience sampling technique based on pre-defined inclusion and exclusion criteria. To test reliability of inter/intra observer of ultimate final Urdu Version of Oxford Knee Score will be filled from patients on the equivalent day, by 2 different bystanders, and for inter observer valuation, with an interval of 30 minutes between the first and second application. Third assessment will be carried out after 7 days of the Observer -1, for intra-observer assessment. Data will be entered and analyzed Cronbach alpha value. Test-retest reliability will be assessed using an intra-class correlation coefficient. Urdu Version of Oxford Knee Score will be evaluated for content validity, construct validity, criterion validity and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed knee Osteoarthritis patients were included
* Both male and female patients were included
* Both unilateral and bilateral knee Osteoarthritis patients were included
* Patients were included who fulfilled the American college of rheumatology criteria
* Patients were included between the age of 35-80 Y old patients

Exclusion Criteria:

* Patients with any heart problem were excluded
* Patients with peripheral vascular injury were excluded

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee Osteoarthritis were included from Pakistan
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
Oxford knee score | day 1
  Oxford knee score is 12 items self-evaluation form which is used to evaluate the knee Osteoarthritis. Oxford knee score is used to evaluate pain and physical disability.
Western Ontario McMaster universities osteoarthritis index | day 1
  Western Ontario McMaster universities osteoarthritis index is a 24 items to evaluate knee Osteoarthritis. First 5 items are used to evaluate pain, 6 and 7 items are used to evaluate stiffness and next 8 to 24 questions are used to access physical function.
International Knee Documentation Committee | day 1
  International Knee Documentation Committee has 19 items. It is used to evaluate knee Osteoarthritis and ligament injuries. The International Knee Documentation Committee is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No